CLINICAL TRIAL: NCT02665559
Title: Transversal Study, Prospective, to Evaluate the Prevalence and Factors Associated With Hypogonadism in HIV + Men
Brief Title: Study of the Prevalence and Associated Factors With Hypogonadism in HIV + Men
Acronym: HYPOG
Status: Completed | Type: Observational
Sponsor: Tourcoing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HYPOGONADISME
Record Dates: First submitted 2013-06-05; First posted 2016-01-27 (Estimated); Last update posted 2018-09-17 (Actual); Status verified 2016-01

CONDITIONS: Hypogonadism; HIV
Keywords: HIV; Hypogonadism; Metabolic Syndrom; Reservoirs; Osteodensitometry; Erectil dysfonction; Depression
MeSH Terms: conditions — Hypogonadism; Depression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — HIV-DNA quantification on PBMCs sample
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Hypogonadism group: a cross-sectional and prospective study, in HIV-infected men less than 50 years old, with HIV-RNA ≤ 50 cop/mL under ART who had never presented AIDS

SUMMARY:
Testosterone deficiency is classically associated with the development of metabolic syndrome, osteoporosis, erectile disorder and / or a reduced libido, a depressive syndrome and alteration of the quality of patients life.

Chronicity of HIV infection leads to several disorders as fever, chronic stress, weight loss and cachexia which are the cause of hypogonadotropic hypogonadism. On the other hand, abnormal secretion of cytokines, secondary to the infection may alter the Leydig cells causing a hypergonadotropic hypogonadism and disrupts steroidogenesis. Cases of testicular invasion by lymphoma or Kaposi's syndromes have also been described.

The advent of antiretroviral therapy has reduced the prevalence of hypogonadism in patients infected with HIV that is currently about 20%. This prevalence remains about 20%, regardless of the antiretroviral therapy and CD4-T cell count.

No study to our knowledge has so far assessed exhaustively the clinical features, biological, therapeutic and paraclinical of hypotestosteronemiae while assessing the level of total serum testosterone, SHBG and serum free testosterone, among HIV infected patients in the European population.

DETAILED DESCRIPTION:
Assess the prevalence and clinical, biological, paraclinical and therapeutic factors associated with primary or secondary hypogonadism in HIV treated and virologically suppressed patients.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18-50 years at the inclusion visit
* Under antiretroviral treatment for more than six months with undetectable viral load (last sample older than four months before the visit of run)
* Infection by HIV-1 positive (confirmation by a full Western blot or by measurement of plasma HIV RNA prior to the inclusion)
* Lack of co-infections HBV, HCV (last negative serology older than 6 months before the screening visit inclusion)
* Consent signed by the patient and the investigator the day of the inclusion and before any examination required by the test (Article L1122-1-1 the Code of Public Health)
* Patient affiliated or beneficiary of a social security system of the European Community member countries (Article L1121-11 of the Code of Public Health).

Exclusion Criteria:

* Infection by HIV-2
* All stages of cirrhosis
* Severe renal impairment (creatinine clearance below 30 ml / min)
* Opportunistic infection during treatment or opportunistic infection in history
* Neoplastic pathology being processed
* Taken in the previous 3 months of testosterone and other anabolic agents, antiandrogens, estrogens, glucocorticoids, analog GnRH, growth hormone or human insulin-like growth factor-1 (IGF-1)
* Pituitary, adrenal or testicular pathologies , treated or not
* Presence or history of psychotic disorder and / or high suicide risk
* Refusal to participate
* No one under safeguard justice
* Patients participating in another research evaluating other treatments and including an exclusion period ongoing at the inclusion

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: HIV-infected men, treated by cART and presenting an undetectable viral load
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2013-01; Primary Completion 2016-06 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Testosteron Level | up to 1 year
  Quantification of testosteron level at Day 0 of the inclusion and at Day 8 after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Antoine CHERET, M.D.,PhD., Study Chair — Tourcoing Hospital; Armelle PASQUET, M.D., Study Director — Tourcoing Hospital
Locations (1):
- Tourcoing Hospital, Tourcoing, France

IPD SHARING:
Plan to Share IPD: Yes
data are reported on a informatic folder centralized at Tourcoing Hospital with anonymous number for each patient Each patient receive by their own practician the biologics data